CLINICAL TRIAL: NCT02813863
Title: The Drug-drug Interaction of SP2086 and Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP2086-104
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SP2086 and Metformin (Experimental): In the first day,the subject takes metformin 1000mg once,and from Day 4 to Day 7 they need to take SP2086 100mg everyday. In Day 8,they will be given SP2086 100mg and metformin 1000mg.
  Interventions: Drug: SP2086; Drug: Metformin

INTERVENTIONS:
Drug: SP2086
Drug: Metformin

SUMMARY:
This is an open single and self-control study,planning to recruit 24 cases of healthy male volunteers.In the study,subjects were given SP2086 and metformin,and collects blood samples before and after medcine.The purpose is to evaluate the drug interaction between SP2086 and Metformin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a body mass index (BMI, a measure of a person's weight in relation to height) between 19 and 26 kg/m2,weight among of 50-100kg.
* willing to using contraception during the study and after the 6 months.

Exclusion Criteria:

* History of diabetes
* History of heart failure or renal insufficiency
* Urinary tract infections, or vulvovaginal mycotic infections
* History of or current clinically significant medical illness as determined by the Investigator
* History of clinically significant allergies, especially known hypersensitivity or intolerance to lactose
* Known allergy to SP2086 or metformin or any of the excipients of the formulation of SP2086 or metformin

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to Day 9
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of metformin
The area under the plasma concentration-time curve (AUC) of SP2086 | up to Day 9
  AUC (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of metformin
The maximum plasma concentration (Cmax) of SP2086 acid | up to Day 9
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of metformin
The area under the plasma concentration-time curve (AUC) of SP2086 acid | up to Day 9
  AUC (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of metformin
The maximum plasma concentration (Cmax) of Metformin | up to Day 9
  Cmax (a measure of the body's exposure to metformin) will be compared. before and after administration of multiple doses of SP2086
The area under the plasma concentration-time curve (AUC) of metformin | up to Day 9
  AUC (a measure of the body's exposure to metformin) will be compared before and after administration of multiple doses of SP2086

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 9